CLINICAL TRIAL: NCT00754663
Title: BETA: Beneficial Effects of Exercise Training in Patients With Implantable Cardioverter-Defibrillators
Brief Title: Exercise Training in Patients With Cardioverter-Defibrillators
Acronym: BETA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Dr. med. Slawomir Weretka, University Hospital Tübingen, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 01
Record Dates: First submitted 2008-08-04; First posted 2008-09-18 (Estimated); Last update posted 2008-09-18 (Estimated); Status verified 2008-09

CONDITIONS: Arrhythmia
Keywords: exercise; implantable cardioverter-defibrillator; arrhythmia
MeSH Terms: conditions — Arrhythmias, Cardiac; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): exercise training
  Interventions: Behavioral: exercise training
- 2 (Placebo Comparator): control arm: normal behavior, no additional exercise will be advised
  Interventions: Behavioral: exercise training

INTERVENTIONS:
Behavioral: exercise training — walking training at least 3 times a week

SUMMARY:
Exercise therapy has proven to be an effective additive therapy in patients with cardiovascular diseases. The prognostic value of physical activity is well established in patients with congestive heart failure. Therefore the investigators assumed that the population of patients with implantable cardioverter-defibrillators (ICD) with impaired left ventricular function may also benefit from a cardiovascular training in terms of improved quality of life and reduction of ventricular arrhythmia. The data on feasibility, risk and therapeutic effects of exercise training are very limited or not available.

This prospective randomized study examines the feasibility and benefits of exercise therapy in patients with ICD and congestive heart failure.

DETAILED DESCRIPTION:
Detailed anamnesis and a clinical examination will be performed in order to determine the patient's eligibility for the study. The randomisation either to the exercise- or to the control-arm will be performed at baseline. Follow-up visits are planned after four weeks and after three months same for both arms. The close-up visit is planned after 6 months.

The exercise-arm starts off with an introduction into physical training at the Department of Sports Medicine at the University in Tübingen. Ergospirometry and 6-min walk test will be performed to determine the patients' performance. Then the patients will be encouraged to exercise at home. The scales and intensities of physical training will vary interpersonally depending on patients individual performance. Pedometers and the ICD-integrated "Cardiac Compass" function will be used to verify work load, intensity and duration of the physical strain. The patients will be consulted by telephone regularly to affirm the study compliance. The physical activity in the control-arm will be monitored using the ICD-integrated "Cardiac Compass" function.

ICD-programming

* VT/SVT discrimination "on",
* "Cardiac Compass" feature "on"
* VT/VF detection and pacing-programming remain adjusted to clinical situation of the patient

Baseline- and follow-up visits

* Anamnesis, NYHA-stadium, patients' demographic data: sex, age, weight, hight, concomitant diseases and current medication
* Clinical examination: weight, inflow-congestion, edema, pulmonary signs of cardiac decompensation
* Chest- x-ray (baseline, 6 moths FU)
* 6-min walk test (baseline, 6 moths FU)
* Blood take (baseline, 6 moths FU) standard examinations including blood morphology, troponin, renal retention parameters, transaminases)
* Determination of the BNP plasma level
* Echocardiography (baseline, 6 moths FU): left-ventricular function (EF) and diameter, valvular function, estimating of systolic pulmonary arterial pressure (PAP sys.).
* Ergospirometry (baseline, 6 moths FU):peak-oxygen-uptake-volume, starting at 10 Watt with increase of the work load 12 Watts per minute until the work load capacity has been reached. The achieved VO2 value is defined as the 100 % oxygen-uptake. At home the patients are supposed to exercise at about 70 % of their VO2 peak.
* Measurement/Recording of the peripheral oxygen-uptake of the muscle with near-infrared-spectroscopy simultaneously with the bicycle-ergometric exposure.
* Complete interrogation of the ICD-memory, acquisition of the "Cardiac-Compass"-data, sensing- and threshold-test, recording of electrical impedance and checking of the battery-status, impedance and checking of the battery-status
* Acquisition of the standardized questionnaires concerning quality-of-life, personality, depression and anxiety: PHQ-D, DS14, FSGV 1.0 and GAD-7.

Definition of adverse event

* Adverse event (AE): Any decrease of existential orientation, unwanted incidence, subjective or objective symptom of any kind of disease, impairment or any accident, that may or may not be connected to the study is defined as an (AE).
* Severe adverse event (SAE): A SAE is an event which is life-threatening or deadly, causes significant or chronic damage, requires hospitalization or threatens the patient's physical inviolability in any other way.

ELIGIBILITY:
Inclusion Criteria:

* both gender at a minimum age of 18 years
* ICD-systems with "Cardiac-Compass" (Medtronic)-diagnostic feature
* ICD system implanted for at least three months
* congestive heart failure, NYHA II and III
* LVEF ≤ 40 %
* compensated state, optimized and stable pharmacological therapy at least for the last three months
* load capacity of at least 50 watt at baseline.

Exclusion Criteria:

* unable or unwilling to give informed consent
* acute coronary syndrome during the past thirty days
* hemodynamically relevant valvular defect
* instable arterial hypertension
* severe COPD
* reduced work load capacity caused by instable angina pectoris, peripheral vascular, neurological or orthopaedic concomitant disease
* hypertrophic obstructive cardiomyopathy (HOCM)
* pulmonary-arterial hypertension (PAP systolic ≥ 60 mmHg).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-09 (Estimated); Study Completion 2009-11 (Estimated)

PRIMARY OUTCOMES:
Reduction of arrhythmia burden, heart rate trend, increase in patients activity. | 6 months

SECONDARY OUTCOMES:
Ineffective ICD-interventions, injury risk due to syncope, hospitalization, death. LVEF (echocardiography), VO2max, anaerobic threshold (AT), respiratory compensation point (RCP) and equivalents for O2 and CO2 (ergospirometry) BNP plasma level | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Slawomir Weretka, MD, Principal Investigator — University Hospital Tuebingen; Juergen Schreieck, MD, Study Chair — University Hospital Tuebingen
Locations (1):
- University Clinic, Dept. of Cardiology, Tübingen, Baden-Wurttemberg, Germany

REFERENCES:
- [Background] Lakka TA, Venalainen JM, Rauramaa R, Salonen R, Tuomilehto J, Salonen JT. Relation of leisure-time physical activity and cardiorespiratory fitness to the risk of acute myocardial infarction. N Engl J Med. 1994 Jun 2;330(22):1549-54. doi: 10.1056/NEJM199406023302201. PMID 8177243
- [Background] Schuler G. [Physical activity]. Z Kardiol. 2005;94 Suppl 3:III/11-4. doi: 10.1007/s00392-005-1303-1. German. PMID 16258787
- [Background] Dursch M, Schulz O. [Restructuring cardiovascular exercise therapy in Germany with reference to current international guidelines]. Herz. 2003 Aug;28(5):349-58. doi: 10.1007/s00059-003-2438-3. German. PMID 12928734
- [Background] Schulz O, Dursch M. [From bench to bicycle. Risk assessment in connection with sports activities and exercise programs in the primary and secondary prevention of cardiovascular diseases]. Herz. 2003 Aug;28(5):359-73. doi: 10.1007/s00059-003-2463-9. German. PMID 12928735
- [Background] Erbs S, Linke A, Gielen S, Fiehn E, Walther C, Yu J, Adams V, Schuler G, Hambrecht R. Exercise training in patients with severe chronic heart failure: impact on left ventricular performance and cardiac size. A retrospective analysis of the Leipzig Heart Failure Training Trial. Eur J Cardiovasc Prev Rehabil. 2003 Oct;10(5):336-44. doi: 10.1097/01.hjr.0000099031.38268.27. PMID 14663295
- [Background] Hambrecht R, Gielen S, Linke A, Fiehn E, Yu J, Walther C, Schoene N, Schuler G. Effects of exercise training on left ventricular function and peripheral resistance in patients with chronic heart failure: A randomized trial. JAMA. 2000 Jun 21;283(23):3095-101. doi: 10.1001/jama.283.23.3095. PMID 10865304
- [Background] Belardinelli R, Georgiou D, Cianci G, Purcaro A. Randomized, controlled trial of long-term moderate exercise training in chronic heart failure: effects on functional capacity, quality of life, and clinical outcome. Circulation. 1999 Mar 9;99(9):1173-82. doi: 10.1161/01.cir.99.9.1173. PMID 10069785
- [Background] Kamke W, Dovifat C, Schranz M, Behrens S, Moesenthin J, Voller H. Cardiac rehabilitation in patients with implantable defibrillators. Feasibility and complications. Z Kardiol. 2003 Oct;92(10):869-75. doi: 10.1007/s00392-003-0997-1. PMID 14579052
- [Background] Vanhees L, Schepers D, Heidbuchel H, Defoor J, Fagard R. Exercise performance and training in patients with implantable cardioverter-defibrillators and coronary heart disease. Am J Cardiol. 2001 Mar 15;87(6):712-5. doi: 10.1016/s0002-9149(00)01488-0. PMID 11249888
- [Background] Vanhees L, Kornaat M, Defoor J, Aufdemkampe G, Schepers D, Stevens A, Van Exel H, Van Den Beld J, Heidbuchel H, Fagard R. Effect of exercise training in patients with an implantable cardioverter defibrillator. Eur Heart J. 2004 Jul;25(13):1120-6. doi: 10.1016/j.ehj.2004.04.034. PMID 15231370
- [Background] Lampert R, Cannom D, Olshansky B. Safety of sports participation in patients with implantable cardioverter defibrillators: a survey of heart rhythm society members. J Cardiovasc Electrophysiol. 2006 Jan;17(1):11-5. doi: 10.1111/j.1540-8167.2005.00331.x. PMID 16426392
- [Background] Hunt SA, Abraham WT, Chin MH, Feldman AM, Francis GS, Ganiats TG, Jessup M, Konstam MA, Mancini DM, Michl K, Oates JA, Rahko PS, Silver MA, Stevenson LW, Yancy CW, Antman EM, Smith SC Jr, Adams CD, Anderson JL, Faxon DP, Fuster V, Halperin JL, Hiratzka LF, Jacobs AK, Nishimura R, Ornato JP, Page RL, Riegel B; American College of Cardiology; American Heart Association Task Force on Practice Guidelines; American College of Chest Physicians; International Society for Heart and Lung Transplantation; Heart Rhythm Society. ACC/AHA 2005 Guideline Update for the Diagnosis and Management of Chronic Heart Failure in the Adult: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Writing Committee to Update the 2001 Guidelines for the Evaluation and Management of Heart Failure): developed in collaboration with the American College of Chest Physicians and the International Society for Heart and Lung Transplantation: endorsed by the Heart Rhythm Society. Circulation. 2005 Sep 20;112(12):e154-235. doi: 10.1161/CIRCULATIONAHA.105.167586. Epub 2005 Sep 13. No abstract available. PMID 16160202
- See also: Study projects/ Dept. of Cardiology Electrophysiology, Univ. Clinic Tübingen — http://www.medizin.uni-tuebingen.de/kardiologie/forschung/frmforsc.htm